CLINICAL TRIAL: NCT02680327
Title: A Feasibility Study on: Advance Care Planning (ACP) in Elderly Cardiac Surgery Patients
Brief Title: Advance Care Planning (ACP) in Elderly Cardiac Surgery Patients
Acronym: DIMAN
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Montreal Heart Institute (Other)
Responsible Party: Principal Investigator, Jennifer Cogan, Associate Professor, MSc, MD, FRCPC,, Montreal Heart Institute
Other Study IDs: ICM 15-1875
Record Dates: First submitted 2016-01-29; First posted 2016-02-11 (Estimated); Last update posted 2016-02-11 (Estimated); Status verified 2016-02

CONDITIONS: Advanced Care Planning

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
This is a prospective epidemiological pilot study to evaluate the feasibility of recruiting and retaining patients in a large multicenter study that will audit Advanced Care Planning (ACP) practices and satisfaction with End Of Life (EOL) communication and decision-making in patients undergoing cardiac surgery using the current validated questionnaires and methodology.

DETAILED DESCRIPTION:
Study Procedures:

Once patients have signed an informed consent they will be asked to complete the ACP evaluation questionnaire. Their level of frailty will be assessed with the 5-meter walk test. Two weeks after discharge (+ or - 7 days) they will be contacted by phone in order to complete 3 sections of the CANHELP questionnaire.

Study Tools

Patient questionnaires:

1. ACP Evaluation questionnaire: 5 questions about advance care planning on admission to hospital from CANHELP study (time predicted 10 minutes)
2. CANHELP questionnaire (sections relationship with doctors, communication and decision making) 2 weeks after discharge (time predicted 25 minutes)

Patient test:

1. 5-minute gait speed

   Patient Assessment Data
2. Standard Demographics
3. Anthropometric data
4. Cardiac variables
5. Comorbidities
6. Lab Values
7. Frailty (assessed using 5-meter gait speed)

Post-surgical outcome data (will be sought in the chart after 30 days post-surgery)

1. Outcome
2. Complications

ELIGIBILITY:
Inclusion Criteria:

* Age and over 70 years
* Admitted for cardiac surgery;
* Able to speak English or French;

Exclusion Criteria:

* Age under 70 years;
* Unable to participate in the follow-up telephone survey;
* Unable to speak English or French.

Ages: 70 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Patients 70 years of age and over admitted for cardiac surgery that requires a general anesthetic (either via median sternotomy, minimally invasive or percutaneous approach);
Sampling Method: Non-Probability Sample
Enrollment: 35 (Estimated)
Dates: Start 2015-10; Primary Completion 2016-04 (Estimated); Study Completion 2016-07 (Estimated)

PRIMARY OUTCOMES:
Successful study completion | 1 month
  To estimate the proportion of patients who successfully completed all the study tasks;
Time frame | 1 month
  To evaluate the time frame required to enroll and complete the study for 35 patients;
Gait test | 1 month
  To evaluate the length of time required perform the gait test (in minutes);
patient retention | 1 month
  To evaluate patient retention (percent of patients who complete the study);
Screen failure rate | 1 month
  To evaluate the screen failure rate

SECONDARY OUTCOMES:
Overall satisfaction | 1 month
  To assess the patient's overall satisfaction with goals of care communication (question 1 of CANHELP questionnaire; (5 point Likert scale));
Prevalence of ACP | 1 month
  To determine, from the perspective of the acutely ill patient, the prevalence of Advanced Care Planning (ACP) directives;
Percentage of frail patients | 1 month
  To evaluate proportion of patients evaluated as frail using the 5-meter walk test;
Level of correlation between "level of frailty" and "satisfaction with decision making". | 1 month
  To evaluate the level of correlation between "satisfaction with decision making" and level of frailty.

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Cogan, MD, FRCPC, Principal Investigator — Montreal Heart Institute
Locations (1):
- Montreal Heart Institute, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Pfisterer M, Buser P, Osswald S, Allemann U, Amann W, Angehrn W, Eeckhout E, Erne P, Estlinbaum W, Kuster G, Moccetti T, Naegeli B, Rickenbacher P; Trial of Invasive versus Medical therapy in Elderly patients (TIME) Investigators. Outcome of elderly patients with chronic symptomatic coronary artery disease with an invasive vs optimized medical treatment strategy: one-year results of the randomized TIME trial. JAMA. 2003 Mar 5;289(9):1117-23. doi: 10.1001/jama.289.9.1117. PMID 12622581
- [Result] Alexander KP, Anstrom KJ, Muhlbaier LH, Grosswald RD, Smith PK, Jones RH, Peterson ED. Outcomes of cardiac surgery in patients > or = 80 years: results from the National Cardiovascular Network. J Am Coll Cardiol. 2000 Mar 1;35(3):731-8. doi: 10.1016/s0735-1097(99)00606-3. PMID 10716477
- [Result] Graham MM, Ghali WA, Faris PD, Galbraith PD, Norris CM, Knudtson ML; Alberta Provincial Project for Outcomes Assessment in Coronary Heart Disease (APPROACH) Investigators. Survival after coronary revascularization in the elderly. Circulation. 2002 May 21;105(20):2378-84. doi: 10.1161/01.cir.0000016640.99114.3d. PMID 12021224
- [Result] Afilalo J, Eisenberg MJ, Morin JF, Bergman H, Monette J, Noiseux N, Perrault LP, Alexander KP, Langlois Y, Dendukuri N, Chamoun P, Kasparian G, Robichaud S, Gharacholou SM, Boivin JF. Gait speed as an incremental predictor of mortality and major morbidity in elderly patients undergoing cardiac surgery. J Am Coll Cardiol. 2010 Nov 9;56(20):1668-76. doi: 10.1016/j.jacc.2010.06.039. PMID 21050978
- [Result] Heyland DK, Barwich D, Pichora D, Dodek P, Lamontagne F, You JJ, Tayler C, Porterfield P, Sinuff T, Simon J; ACCEPT (Advance Care Planning Evaluation in Elderly Patients) Study Team; Canadian Researchers at the End of Life Network (CARENET). Failure to engage hospitalized elderly patients and their families in advance care planning. JAMA Intern Med. 2013 May 13;173(9):778-87. doi: 10.1001/jamainternmed.2013.180. PMID 23545563
- [Result] Ehlenbach WJ, Barnato AE, Curtis JR, Kreuter W, Koepsell TD, Deyo RA, Stapleton RD. Epidemiologic study of in-hospital cardiopulmonary resuscitation in the elderly. N Engl J Med. 2009 Jul 2;361(1):22-31. doi: 10.1056/NEJMoa0810245. PMID 19571280
- [Result] Wright AA, Zhang B, Ray A, Mack JW, Trice E, Balboni T, Mitchell SL, Jackson VA, Block SD, Maciejewski PK, Prigerson HG. Associations between end-of-life discussions, patient mental health, medical care near death, and caregiver bereavement adjustment. JAMA. 2008 Oct 8;300(14):1665-73. doi: 10.1001/jama.300.14.1665. PMID 18840840
- [Result] You JJ, Fowler RA, Heyland DK; Canadian Researchers at the End of Life Network (CARENET). Just ask: discussing goals of care with patients in hospital with serious illness. CMAJ. 2014 Apr 1;186(6):425-32. doi: 10.1503/cmaj.121274. Epub 2013 Jul 15. No abstract available. PMID 23857860
- [Result] Heyland DK, Cook DJ, Rocker GM, Dodek PM, Kutsogiannis DJ, Skrobik Y, Jiang X, Day AG, Cohen SR; Canadian Researchers at the End of Life Network. The development and validation of a novel questionnaire to measure patient and family satisfaction with end-of-life care: the Canadian Health Care Evaluation Project (CANHELP) Questionnaire. Palliat Med. 2010 Oct;24(7):682-95. doi: 10.1177/0269216310373168. Epub 2010 Jul 6. PMID 20605850
- [Result] Heyland DK, Cook DJ, Rocker GM, Dodek PM, Kutsogiannis DJ, Skrobik Y, Jiang X, Day AG, Cohen SR; Canadian Researchers at the End of Life Network (CARENET). Defining priorities for improving end-of-life care in Canada. CMAJ. 2010 Nov 9;182(16):E747-52. doi: 10.1503/cmaj.100131. Epub 2010 Oct 4. PMID 20921249
- [Result] Purser JL, Kuchibhatla MN, Fillenbaum GG, Harding T, Peterson ED, Alexander KP. Identifying frailty in hospitalized older adults with significant coronary artery disease. J Am Geriatr Soc. 2006 Nov;54(11):1674-81. doi: 10.1111/j.1532-5415.2006.00914.x. PMID 17087693
- [Result] Cesari M, Kritchevsky SB, Penninx BW, Nicklas BJ, Simonsick EM, Newman AB, Tylavsky FA, Brach JS, Satterfield S, Bauer DC, Visser M, Rubin SM, Harris TB, Pahor M. Prognostic value of usual gait speed in well-functioning older people--results from the Health, Aging and Body Composition Study. J Am Geriatr Soc. 2005 Oct;53(10):1675-80. doi: 10.1111/j.1532-5415.2005.53501.x. PMID 16181165
- [Result] Dumurgier J, Elbaz A, Ducimetiere P, Tavernier B, Alperovitch A, Tzourio C. Slow walking speed and cardiovascular death in well functioning older adults: prospective cohort study. BMJ. 2009 Nov 10;339:b4460. doi: 10.1136/bmj.b4460. PMID 19903980